CLINICAL TRIAL: NCT07115966
Title: Impact of a Simple Automated Best Practice Alert (BPA) on Quantity and Quality of In-hospital Antibiotic Use - a Stepped-wedge, Cluster Randomized, Controlled Trial
Brief Title: Impact of a Simple Automated Best Practice Alert (BPA) on Quantity and Quality of In-hospital Antibiotic Use in a Tertiary and Three Secondary Hospitals
Acronym: TARGET
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Prevention
Other Study IDs: 2025-00735
Record Dates: First submitted 2025-08-04; First posted 2025-08-11 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Antibiotic Prescriptions; In-Patient Treatment
Keywords: best practice alert; quanlity and quantity of antibiotic use; in-patients

STUDY DESIGN:
Intervention Model Description: Wards will be cluster-randomized according to specialty and antibiotic use (DASC/PA), based on retrospective data. The BPA will be activated in a stepwise manner for each cluster every two months over a 12-month period. By the end of the study, the BPA will be active in all participating wards.
Who Masked: Outcomes Assessor
Masking Description: Cluster allocation will also be blinded to the wards and prescribers; however, prescribers may become aware of their cluster assignment when working across different wards in both intervention and control clusters, based on whether or not they receive the BPA.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Best practice alert (BPA) (Experimental): Intervention:
  The BPA will appear to the prescribing physician for every patient on the respective ward.
  Activation of the BPA is ward-based.
  A total of 58 wards will be stratified according to their focus-surgical, medical, intermediate care, rehabilitation, or pediatric-and grouped based on their baseline antibiotic consumption, measured in days of antibiotic spectrum coverage per patient admission (DASC/PA). This stratification will result in 9 to 10 clusters across 6 groups.
  The clusters will then be randomized to the timing of BPA activation, and all wards will sequentially switch to the BPA arm every 2 months over a 12-month period.
  By the end of the trial, after 12 months, all wards will be using the automated BPA.
  Interventions: Behavioral: Computerized decision support by best practice alert (BPA)
- Controls - No BPA (No Intervention): Control: standard patient care with no BPA activated. By the end of the trial, after 12 months, all wards will be using the automated BPA.

INTERVENTIONS:
Behavioral: Computerized decision support by best practice alert (BPA) — The antimicrobial stewardship intervention encourages prescribers by a simple alert to follow guidelines for reviewing antimicrobial prescriptions after a set timeframe for potential de-escalation to targeted therapy or discontinuation of the antibiotics, as recommended by national and international guidelines.
  An automated simple BPA will trigger after an antibiotic prescription with therapeutic indication (72 hours) or surgical prophylaxis (24 hours, reminding prescribers to reassess treatment for possible de-escalation, adaption to targeted therapy, or cessation.
  If ignored, the prescription remains unchanged, but the alert will continue until addressed. Prescribers must select reasons for not changing the prescription, such as pending microbiology results. The control group corresponds to the inpatient wards not yet receiving the BPA, where antibiotics are managed according to "standard-of-care".
  Arms: Best practice alert (BPA)

SUMMARY:
The goal of the stepped-wedge cluster-randomized trial is to assess the impact of an antimicrobial stewardship intervention: a simple, automated Best Practice Alert (BPA) that reminds prescribers to reevaluate antibiotic therapy after 72 hours (or 24 hours for prophylaxis), in accordance with guideline recommendations. The primary hypothesis is that this simple BPA reduces antibiotic use in terms of quantity (amount and duration) and quality (spectrum breadth), measured by days of antibiotic spectrum coverage at the patient level (primary outcome), as well as at both patient and cluster levels using various metrics of antibiotic use. The trial will introduce the BPA in a stepwise manner, with all wards implementing it by the end. It will compare the intervention period to the baseline (pre-intervention) and control periods.

ELIGIBILITY:
Inclusion Criteria:

• All inpatient wards with at least 50 PA/year, except those listed in the exclusion criteria

Exclusion Criteria:

Ward level:

* Emergency departments
* Outpatient clinics
* Haemato-oncologic stem cell transplant wards, where daily ID visits are performed
* ICU wards, where daily ID visits are performed

Indvidual patient data for analysis

• Refusal of institutional general consent for further use of patient data

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2025-08-01 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Days of antibiotic spectrum coverage (DASC) per patient admission (PA) | 12 months
  Overall score of days of antibiotic spectrum coverage per patient admission. The score is composed of the breadth of the bacterial spectrum covered by the administered antibiotic (according to Kakiuchi 2022 - the broader the antibiotic spectrum, the higher the score), summed over the number of days the antibiotic is given. Accordingly, there are no maximum or minimum values

SECONDARY OUTCOMES:
Days of antibiotic spectrum coverage (DASC) per patient antibiotic day (PAD) | 12 months
  Overall score of antibiotic spectrum coverage per patient antibiotic day. The score is composed of the breadth of the bacterial spectrum covered by the administered antibiotic (according to Kakiuchi 2022 - the broader the antibiotic spectrum, the higher the score), summed over the number of days the antibiotic is given. Accordingly, there are no maximum or minimum values.
Days of treatment (DOT) per 100 patient days (PD) and per patient admission on ward level | 12 months
  Overall days of treatment (DOT) per 100 patient days (PD) and per patient admission (PA) on ward level
Defined daily doses (DDD) per 100 patient days (PD) and per patient admission (PA) | 12 months
  Overall defined daily doses) per 100 patient days (PD) and per patient admission (PA) on ward level. Standard metrics recommended by WHO for international benchmarking.
Antibiotic (AB) days per patient admission (PA) | 12 months
  No of days an AB per PA gives the proportion of days antibiotics have been applicated, irrespective of single, double, triple combinations, in relation to total PA
In hospital mortality | 12 months
  All cause in hospital mortality
Hospital length of stay (LOS) | 12 months
Unplanned readmission within first 30 days after discharge | 12 months
Patient admission to IMC/ICU from studied wards | 12 months
  Number and proportion of patient admissions to IMC/ICU from studied wards
Number of Infectious diseases (ID) consultation per patient admission (PA) | 12 months
In hospital C. difficile infection incidence within hospital stay per patient admission (PA) and per 100 patient days (PD) | 12 months
Inhospital incidence of multi-drug-resistant-organisms (MDRO) detection per100 patient days (PD) or per patient admission (PA) | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Philipp Jent, PD, Study Chair — Inselgruppe Bern; Nasstasja Wassilew, Dr. med., Principal Investigator — Inselgruppe Bern
Locations (1):
- Inselgruppe, Bern, Switzerland

IPD SHARING:
Plan to Share IPD: No